CLINICAL TRIAL: NCT05911490
Title: Effects of Breaking Prolonged Sitting on 24-h Human Behaviours, Self-feelings, Metabolic Health and Cognition in Healthy Adults
Brief Title: Effects of Breaking Sitting on Human Behaviour and Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Collaborators: Division of Endocrinology and Metabolism, Tri-Service General Hospital (Unknown)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2-108-05-151
Record Dates: First submitted 2023-05-20; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Energy Balance; Physical Activity Level; Cognition; Metabolic Health
Keywords: Breaking up sitting; Eating behaviour; Spontaneous physical activity; Executive function; Energy balance
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged sitting (Active Comparator): Participants sat on a chair during the trial in the laboratory.
  Interventions: Behavioral: Prolonged sitting
- Breaking prolonged sitting (Experimental): Participants walked regularly during the trial in the laboratory.
  Interventions: Behavioral: Breaking prolonged sitting

INTERVENTIONS:
Behavioral: Prolonged sitting — In the laboratory, after consuming 1st meal, participants sat on a chair for 180 min. After 180 min, the 2nd meal was provided. After finishing the 2nd meal, participants sat on a chair for another 120 min. After data collection was completed in the laboratory, participants were asked to keep wearing the same pedometer and to record any food and liquid consumption for the rest of the day (until midnight) under free-living conditions.
  Arms: Prolonged sitting
Behavioral: Breaking prolonged sitting — In the laboratory, after consuming 1st meal, participants walked 2 min on a treadmill every 20 minutes for the following 180 min. For the remainder of the time participants sat on the chair. After 180 min, the 2nd meal was provided. After finishing the 2nd meal, participants continued 2 min of walking every 20 min for the following 120 min. After data collection was completed in the laboratory, participants were asked to keep wearing the same pedometer and to record any food and liquid consumption for the rest of the day (until midnight) under free-living conditions.
  Arms: Breaking prolonged sitting

SUMMARY:
This study primarily aimed to investigate effects of breaking up prolonged sitting with intermittent brisk walking in healthy young individuals on (1) post-trial human behaviours including energy intake and physical activity under free-living conditions and (2) cognitive performance in a simulated workplace environment.

ELIGIBILITY:
Inclusion Criteria:

* Without current and any history of brain injury, neurological disorder, cardiometabolic related diseases, diabetes or cancers.
* Weight stable (not self-reported weight change ± 3 kg at least 3 months)
* Body mass index (BMI) ranging between 18.5 to 27 kg/m2
* Can walk safely on a treadmill

Exclusion Criteria:

* Smokers, post-menopausal female, and volunteers who used any medications that could influence metabolic and inflammatory responses.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Physical activity level | 480 minutes
  Changes in physical activity level (steps) in the free-living conditions
Energy intake | 480 minutes
  Changes in energy intake (kcal) in the free-living conditions
Cognitive performance | 320 minutes
  Changes in cognitive performance (% changes in accuracy) including Task Switching and Flanker tasks
Cognitive function | 320 minutes
  Changes in cognitive performance (% changes in reaction time) Task Switching and Flanker tasks

SECONDARY OUTCOMES:
Postprandial glucose concentrations | 320 minutes
  Changes in postprandial finger pricking glucose concentrations
Blood pressure | 320 minutes
  Changes in systolic blood pressure and diastolic blood pressure
Visual analogue scale (VAS) | 320 minutes
  Changes in self-perceived sensations including appetite, energy and mood (score from 0-100)
Continuous glucose monitoring | 320 minutes
  Changes in different depots of adipose tissue interstitial glucose concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No